CLINICAL TRIAL: NCT04677959
Title: CONNected Electronic Inhalers Asthma Control Trial 2 ("CONNECT 2"), a 24-Week Treatment, Multicenter, Open-Label, Randomized, Parallel Group Comparison, Feasibility Study of Standard of Care Treatment Versus the eMDPI Digital System, to Optimize Outcomes in Patients at Least 13 Years of Age or Older With Asthma
Brief Title: A 24-Week Treatment Study to Compare Standard of Care Versus the eMDPI DS in Participants 13 Years or Older With Asthma
Acronym: CONNECT2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSS-AS-40139
Record Dates: First submitted 2020-12-11; First posted 2020-12-21 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Digital System (DS) (Experimental): DS group participants utilizing the eMDPI DS, including inhaler, smart device application (App), DHP (Cloud solution), and dashboard
  Interventions: Drug: Fluticasone propionate/salmeterol (FS); Drug: Albuterol
- Standard of Care (SoC) Group (Active Comparator): SoC group participants will be treated with their standard of care medications
  Interventions: Drug: Standard of Care Asthma Medication; Drug: Standard of Care Rescue Medication

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol (FS) — FS administered via electronic multidose dry powder inhaler (eMDPI) Digital System (DS) with component devices including smart device application (App), Digital Health Platform (DHP), and provider-facing dashboard
  Arms: Digital System (DS)
Drug: Albuterol — Albuterol administered via electronic multidose dry powder inhaler (eMDPI) Digital System (DS) with component devices including smart device application (App), Digital Health Platform (DHP), and provider-facing dashboard
  Arms: Digital System (DS)
Drug: Standard of Care Asthma Medication — Current inhaled corticosteroid(ICS)/Long-acting beta agonist(LABA) and any additional controller medication for asthma
  Arms: Standard of Care (SoC) Group
Drug: Standard of Care Rescue Medication — Current rescue medication
  Arms: Standard of Care (SoC) Group

SUMMARY:
The primary objective of this study is to demonstrate the effectiveness of the Digital System (DS) in improving asthma control compared to the Standard of Care (SoC) group.

The secondary objective is to describe the asthma management actions by investigational center health care providers (iHCPs) for all participants in both groups, to evaluate short-acting beta2 agonist (SABA) usage and the number of SABA-free days in the DS group, to evaluate adherence patterns to maintenance treatment (FS eMDPI) in the DS group, to assess behavioral correlates of responsiveness to digital health technology among participants for all participants in both groups, to evaluate work productivity and activity impairment in asthma participants in both groups, to assess the usability and acceptability of the DS by participants in the DS group and the investigational center personnel, and to evaluate the safety of FS eMDPI and Albuterol eMDPI.

DETAILED DESCRIPTION:
Study duration will be approximately 27 weeks including a one-week screening period, 24 week treatment period, and a 2 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a documented diagnosis of asthma established at the investigational center at the time of informed consent or the investigator confirms a diagnosis of asthma.
* The participant is currently on treatment with a moderate- to high-dose inhaled corticosteroid (ICS) with long-acting beta agonist (LABA).
* The participant has an Asthma Control Test score of less than 19 at the screening or baseline visit.
* The participant is willing to discontinue all other maintenance ICS with LABA medications and rescue medications and replace them with the study-provided fluticasone propionate/salmeterol (FS) multidose dry powder inhaler with integrated electronic module (eMDPI) and Albuterol eMDPI, respectively, for the duration of the trial, if randomized to the Digital System group. All other asthma maintenance medications, except for ICS with LABA, may be continued.

  * Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* The participant is currently being treated prior to enrollment with a digital inhaler system, including the Digihaler system or an external "bolt on" digital system designed to monitor inhaler usage, such as the Propeller Health or Adherium systems.
* The participant has any clinically significant uncontrolled medical condition (treated or untreated) other than asthma, which in the view of the investigator would preclude participation.
* The participant was hospitalized for severe asthma in the last 30 days.
* The participant has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the patient's ability to participate in this study.

  * Additional criteria apply, please contact the investigator for more information.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (46):
- United States (46):
  - Teva Investigational Site 14971, Phoenix, Arizona
  - Teva Investigational Site 14974, Fountain Valley, California
  - Teva Investigational Site 14982, Los Angeles, California
  - Teva Investigational Site 14945, San Diego, California
  - Teva Investigational Site 14946, San Diego, California
  - Teva Investigational Site 14966, Colorado Springs, Colorado
  - Teva Investigational Site 14962, Wheat Ridge, Colorado
  - Teva Investigational Site 14943, Aventura, Florida
  - Teva Investigational Site 14969, Boynton Beach, Florida
  - Teva Investigational Site 14978, Cutler Bay, Florida
  - Teva Investigational Site 14955, Fort Lauderdale, Florida
  - Teva Investigational Site 14984, Hialeah, Florida
  - Teva Investigational Site 14979, Hialeah, Florida
  - Teva Investigational Site 14953, Miami, Florida
  - Teva Investigational Site 14975, Miami, Florida
  - Teva Investigational Site 14944, Miami, Florida
  - Teva Investigational Site 14970, Miami, Florida
  - Teva Investigational Site 14960, Miami Lakes, Florida
  - Teva Investigational Site 14981, Sarasota, Florida
  - Teva Investigational Site 14951, Tallahassee, Florida
  - Teva Investigational Site 14942, Savannah, Georgia
  - Teva Investigational Site 14947, Boise, Idaho
  - Teva Investigational Site 14961, Glenview, Illinois
  - Teva Investigational Site 14972, Springfield, Illinois
  - Teva Investigational Site 14950, Lexington, Kentucky
  - Teva Investigational Site 14949, Owensboro, Kentucky
  - Teva Investigational Site 14976, Bangor, Maine
  - Teva Investigational Site 14983, White Marsh, Maryland
  - Teva Investigational Site 14964, Farmington Hills, Michigan
  - Teva Investigational Site 14990, Bellevue, Nebraska
  - Teva Investigational Site 14977, Lincoln, Nebraska
  - Teva Investigational Site 14957, Toms River, New Jersey
  - Teva Investigational Site 14956, Hollis, New York
  - Teva Investigational Site 14954, Gastonia, North Carolina
  - Teva Investigational Site 14941, Cincinnati, Ohio
  - Teva Investigational Site 14968, Toledo, Ohio
  - Teva Investigational Site 14952, Oklahoma City, Oklahoma
  - Teva Investigational Site 14958, Oklahoma City, Oklahoma
  - Teva Investigational Site 14967, Pittsburgh, Pennsylvania
  - Teva Investigational Site 14988, Providence, Rhode Island
  - Teva Investigational Site 14989, North Charleston, South Carolina
  - Teva Investigational Site 14985, Boerne, Texas
  - Teva Investigational Site 14963, Houston, Texas
  - Teva Investigational Site 14948, Waco, Texas
  - Teva Investigational Site 14987, Draper, Utah
  - Teva Investigational Site 14965, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SoC): Participants were treated with their current SoC treatment and did not use the digital system during the treatment period. Participants were reimbursed or given a voucher to use to purchase their existing maintenance inhaled corticosteroid (ICS)/ long acting beta2 agonist (LABA) and short-acting beta2 agonist (SABA) inhalers and reliever medications.
- Digital System (DS): Participants were trained on the use of the multidose dry powder inhaler with integrated electronic module (eMDPI) DS (including instructions on how to use both the eMDPI and the App) and, upon demonstrating competency, participants had their maintenance ICS/LABA and SABA inhalers switched to the fluticasone propionate/salmeterol (FS) eMDPI (at a dose of fluticasone comparable to their most recent current ICS dose) and their reliever treatment switched to the albuterol eMDPI. The eMDPI DS consisted of 4 devices: Device 1: albuterol/FS eMDPI (the test investigational medicinal product [IMP]); Device 2: Patient-facing smart device App; Device 3: Digital health platform (DHP) (Cloud solution); and Device 4: Provider-facing Dashboard. Participants received albuterol 1 to 2 oral inhalations every 4 to 6 hours, as needed or FS 1 oral inhalation twice daily for 24 weeks.
Period: Overall Study
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Started | 185 | 242
Safety Analysis Set (All participants in the DS group who received at least 1 dose of IMP and all participants in the SoC group.) | 185 | 224
Completed | 173 | 183
Not Completed | 12 | 59
Not completed — Adverse Event | 1 | 9
Not completed — Withdrawal by Subject | 2 | 15
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Non-compliance with study drug | 0 | 2
Not completed — Protocol deviation | 0 | 11
Not completed — Lost to Follow-up | 9 | 13
Not completed — Other than specified | 0 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Standard of Care (SoC): Participants were treated with their current SoC treatment and did not use the digital system during the treatment period. Participants were reimbursed or given a voucher to use to purchase their existing maintenance ICS/ LABA and SABA inhalers and reliever medications.
- Digital System (DS): Participants were trained on the use of the multidose dry powder inhaler with eMDPI DS (including instructions on how to use both the eMDPI and the App) and, upon demonstrating competency, participants had their maintenance ICS/LABA and SABA inhalers switched to the FS eMDPI (at a dose of fluticasone comparable to their most recent current ICS dose) and their reliever treatment switched to the albuterol eMDPI. The eMDPI DS consisted of 4 devices: Device 1: albuterol/FS eMDPI (the test IMP); Device 2: Patient-facing smart device App; Device 3: DHP (Cloud solution); and Device 4: Provider-facing Dashboard. Participants received albuterol 1 to 2 oral inhalations every 4 to 6 hours, as needed or FS 1 oral inhalation twice daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | Digital System (DS) | Total
Number analyzed (Participants) | 185 | 242 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (17.72) | 46.9 (18.36) | 46.8 (18.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 177 | 293
  Male | 69 | 65 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 80 | 143
  Not Hispanic or Latino | 114 | 157 | 271
  Unknown or Not Reported | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 136 | 185 | 321
  Black or African American | 37 | 45 | 82
  Asian | 7 | 6 | 13
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  Not reported | 2 | 4 | 6
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Well-Controlled Asthma or Reaching Clinically Important Improvement in Asthma Control
Description: A well-controlled asthma was defined as an Asthma Control Test (ACT) score of greater than or equal to 20. Clinically important improvement in asthma control was defined by an increase of at least 3 ACT units from baseline. The ACT was a simple, participant-completed tool used for the assessment of overall asthma control. The ACT included 5 items that assessed daytime and nighttime asthma symptoms, use of reliever medication, and impact of asthma on daily functioning. Each item in the ACT was scored on a 5-point scale ranging from 1 (poor control of asthma) to 5 (well control of asthma), with summation of all items providing scores ranging from 5 to 25. The scores span the continuum of poor control of asthma (score of 5) to complete control of asthma (score of 25), with a cutoff score of 19 and below indicating participants with poorly controlled asthma.
Time Frame: Week 24
Population: The modified intent-to-treat (mITT) analysis set all randomized participants who received at least 1 dose of IMP (IMP was either FS eMDPI or Albuterol eMDPI for the DS group or SoC medication for the SoC group) and at least 1 postbaseline ACT assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 181 | 210
Participants | 112 | 134
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs Digital System (DS); The 95% credible intervals of the odds ratio from the posterior distributions were calculated and presented; Test type: Other; Odds Ratio (OR) = 1.35

2. Secondary Outcome: Number of Discussions Between Participant and Investigational Center Healthcare Professional (iHCP) Regarding Inhaler Technique or Adherence
Description: Number of participants who had discussions with iHCP regarding inhaler technique or adherence are reported.
Time Frame: Baseline up to Week 24
Population: The mITT analysis set all randomized participants who received at least 1 dose of IMP (IMP was either FS eMDPI or Albuterol eMDPI for the DS group or SoC medication for the SoC group) and at least 1 postbaseline ACT assessment. Here 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  0 discussion | 90 | 55
  1 discussion | 33 | 38
  2 discussions | 50 | 55
  3 discussions | 4 | 9
  4 discussions | 0 | 14
  5 discussions | 1 | 4
  6 discussions | 0 | 4
  7 discussions | 0 | 1
  8 discussions | 0 | 6
  10 discussions | 0 | 5
  12 discussions | 0 | 2
  13 discussions | 0 | 1
  14 discussions | 0 | 1
  15 discussions | 0 | 1
  16 discussions | 0 | 1
  17 discussions | 0 | 1
  18 discussions | 0 | 1
  19 discussions | 0 | 4
  20 discussions | 0 | 1
  21 discussions | 0 | 2
  22 discussions | 0 | 1
  23 discussions | 0 | 1
  26 discussions | 0 | 1
  29 discussions | 0 | 1

3. Secondary Outcome: Number of Decreased Doses of Inhaled Medication
Description: Number of participants who received decreased dose of inhaled medication during the 24-week treatment period are reported.
Time Frame: Baseline up to Week 24
Population: The mITT analysis set all randomized participants who received at least 1 dose of IMP (IMP was either FS eMDPI or Albuterol eMDPI for the DS group or SoC medication for the SoC group) and at least 1 postbaseline ACT assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 181 | 210
Participants | 0 | 0

4. Secondary Outcome: Number of Increased Doses of Inhaled Medication
Description: Number of participants who received increased dose of inhaled medication during the 24-week treatment period are reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  No increased doses | 173 | 200
  1 increased dose | 5 | 10

5. Secondary Outcome: Number of Changes to Different Inhaled Medication
Description: Number of participants who received different inhaled medication during the 24-week treatment period are reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  No change to different inhaled medication | 175 | 187
  1 change to different inhaled medication | 3 | 23

6. Secondary Outcome: Number of Additional Inhaled Medication
Description: Number of participants who received additional inhaled medication during the 24-week treatment period are reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  No additional inhaled medication | 173 | 206
  1 additional inhaled medication | 4 | 4
  2 additional inhaled medications | 1 | 0

7. Secondary Outcome: Number of Addition of a Systemic Corticosteroid Medication for Asthma Therapy
Description: Number of participants who received additional systemic corticosteroid medication for asthma therapy during the 24-week treatment period are reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  No addition of a systemic corticosteroid medication for asthma therapy | 173 | 201
  1 addition of a systemic corticosteroid medication for asthma therapy | 3 | 7
  2 addition of a systemic corticosteroid medications for asthma therapy | 0 | 1
  3 addition of a systemic corticosteroid medications for asthma therapy | 2 | 1

8. Secondary Outcome: Frequency of Intervention to Manage Comorbid Conditions Associated With Poor Asthma Control
Description: Number of participants with different frequency of intervention to manage comorbid conditions such as Gastroesophageal Reflux Disease (GERD) and Sinusitis are reported.
Time Frame: Baseline up to Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 178 | 210
Participants
  No intervention to manage comorbid conditions | 169 | 199
  Interventions taken 1 time to manage comorbid conditions | 7 | 7
  Interventions taken 2 times to manage comorbid conditions | 2 | 4

9. Secondary Outcome: Change From Baseline in Mean Weekly SABA Usage at Week 24 for the DS Group
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrograms (μg)
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 158
micrograms (μg) | -12.26 (59.199)

10. Secondary Outcome: Change From Baseline in the Number of SABA-free Days at Week 24 for the DS Group
Description: Number of days a participant did not use the rescue medication in a week are reported.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 158
days | 0.4 (1.94)

11. Secondary Outcome: Change From Baseline in Adherence to Maintenance Treatment (FS eMDPI) at Week 24 for the DS Group
Description: Adherence to maintenance treatment was defined as the percentage of actual inhalation doses taken out of the total number of inhalation doses prescribed over the 24- week treatment period.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of inhalation
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 179
percentage of inhalation | -10.87 (31.717)

12. Secondary Outcome: Change From Baseline in Beliefs About Medicines Questionnaire (BMQ) Concern Subscale Score at Week 24
Description: The BMQ was used to assess cognitive representations of medicine. The Beliefs About Medicines Questionnaire-Specific 11 (BMQ-S11) was an 11-item questionnaire that assessed the representation of medication prescribed for personal use and the BMQ-General assesses beliefs about medicines in general. BMQ concern is a 6-item scale assessing participant's concerns about potential adverse consequences (range: 1=strongly disagree to 5=strongly agree). Participants indicated their degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by the total number of items and multiplied by 5 to give a total score ranging from 5 to 25 (higher scores=stronger beliefs).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 160 | 168
units on a scale | -0.8 (3.34) | -0.9 (4.06)

13. Secondary Outcome: Change From Baseline in BMQ Necessity Subscale Score at Week 24
Description: The BMQ was used to assess cognitive representations of medicine. The Beliefs About Medicines Questionnaire-Specific 11 (BMQ-S11) was an 11-item questionnaire that assessed the representation of medication prescribed for personal use and the BMQ-General assesses beliefs about medicines in general. BMQ necessity is a 5-item scale assessing participant's beliefs about necessity of medications for controlling disease. Participants indicated degree of agreement on a 5-point scale, ranging from 1=strongly disagree to 5=strongly agree. Scores obtained for individual items were summed, divided by the total number of items and multiplied by 5 to give a total score ranging from 5 to 25 (higher scores=stronger beliefs).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 160 | 168
units on a scale | -0.4 (3.27) | -1.3 (3.86)

14. Secondary Outcome: Change From Baseline in Brief Illness Perception Questionnaire (BIPQ) Illness Comprehensibility Subscale Score at Week 24
Description: The BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. Only one item assesses illness comprehensibility or coherence of illness (Item 7: How well do you feel you understand your illness?). This item was rated using a 0 (do not understand at all) to 10 (understand very clearly) response scale. A higher score indicates a stronger illness comprehensibility.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 160 | 168
units on a scale | -0.0 (1.65) | 0.1 (2.04)

15. Secondary Outcome: Change From Baseline in BIPQ Cognitive Subscale Score at Week 24
Description: BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. It comprised 5 items on cognitive representation of illness perception: consequences (Item 1: How much does your illness affect your life? Response range 0 [no affect] - 10 [severe affect]), timeline (Item 2: How long do you think your illness will continue? Response range 0 [a very short time] - 10 [forever]), personal control (Item 3: How much control do you feel you have over your illness? Response range 0 [no control] - 10 [extreme amount of control]), treatment control (Item 4: How much do you think your treatment can help your illness? Response range 0 [not at all] - 10 [extremely helpful]), and identity (Item 5: How much do you experience symptoms from your illness? Response range 0 [no symptoms] - 10 [severe symptoms]). Total BIPQ Cognitive Subscale Score was the sum of all item score and ranged from 0 to 50. A higher score indicates stronger illness perception.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 160 | 168
units on a scale | -2.5 (5.51) | -3.3 (6.83)

16. Secondary Outcome: Change From Baseline in BIPQ Emotional Representations Subscale Score at Week 24
Description: BIPQ was a 9-item questionnaire designed to rapidly assess cognitive and emotional representations of illness. It comprised 2 items on emotional representation: concern (Item 6: How concerned are you about your illness? Response range 0 [not at all concerned] - 10 [extremely concerned]) and emotions (Item 8: How much does your illness affect you emotionally; for example, does it make you angry, scared, upset or depressed? Response range 0 [not at all affected emotionally] - 10 [extremely affected emotionally]). Total BIPQ Emotional Subscale Score was the sum of above 2 items score and ranged from 0 to 20. A higher score indicates extreme emotional representation.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 160 | 168
units on a scale | -1.1 (4.01) | -1.3 (3.98)

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Asthma Questionnaire Score at Week 24
Description: WPAI-asthma is a self-administered instrument to measure asthma-specific performance impairment of work and regular daily activity within the last 7 days and yields 4 types of scores: work time missed (absenteeism), impairment while working (presenteeism or reduced on-the-job effectiveness), overall work impairment (WI) (work productivity loss or absenteeism plus presenteeism) and activity impairment (daily activity impairment). Total score and each score ranged from 0 (not affected/no impairment) to 100 (completely affected/impaired). Higher scores indicated greater impairment and less productivity.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 156 | 167
units on a scale
  Absenteeism: number analyzed (Participants) | 85 | 87
  Absenteeism | -3.56 (14.38) | -0.05 (8.61)
  Presenteeism: number analyzed (Participants) | 92 | 92
  Presenteeism | -10.98 (24.50) | -10.43 (18.57)
  Work productivity loss: number analyzed (Participants) | 85 | 87
  Work productivity loss | -12.18 (26.25) | -9.87 (19.16)
  Activity impairment | -11.22 (23.81) | -15.33 (21.48)

18. Secondary Outcome: System Usability Scale (SUS) Overall Score for DS Group
Description: The SUS was used to explore device acceptability and usability for participants in the DS group. It covered a variety of aspects of system usability, such as the need for support, training, and complexity, and thus giving a global view of subjective assessments of usability. It was a 10-question tool (with five response options; from 1=strongly disagree to 5=strongly agree) that provided a composite measure, ranging from 0 to 100, of the overall usability of the system being studied. Higher scores represent better usability level for the tool.
Time Frame: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital System (DS)
Number analyzed (Participants) | 171
units on a scale
  SUS Overall Score (completed by participants) | 70.0 (19.10)
  Site SUS Overall Score (completed by site): number analyzed (Participants) | 37
  Site SUS Overall Score (completed by site) | 73.2 (18.03)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'. Number of participants with any AEs, and device-related AEs has been reported.
Time Frame: Baseline up to Week 26
Population: The safety analysis set included all participants in the DS group who received at least 1 dose of IMP and all participants in the SoC group.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) | Digital System (DS)
Number analyzed (Participants) | 185 | 224
Participants
  Any AEs | 56 | 77
  Device-related AEs | 0 | 3

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Description: The safety analysis set included all participants in the DS group who received at least 1 dose of IMP and all participants in the SoC group.
Arm/Group | Standard of Care (SoC) | Digital System (DS)
All-Cause Mortality (participants affected / at risk) | 0/185 | 0/224
Serious Adverse Events (participants affected / at risk) | 4/185 | 6/224
Other Adverse Events (participants affected / at risk) | 23/185 | 24/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=185) | Digital System (DS) (N=224)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometrial cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=185) | Digital System (DS) (N=224)
COVID-19 (Infections and infestations) | 15 (16) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 18 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT04677959/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT04677959/SAP_001.pdf